CLINICAL TRIAL: NCT00304278
Title: Phase II Study of RADPLAT and Tarceva in Locally Advanced Head and Neck Squamous Cell Carcinoma (SCCA)
Brief Title: Study of RADPLAT and Tarceva in Locally Advanced Head and Neck Squamous Cell Carcinoma (SCCA)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Southern Illinois University (Other)
Collaborators: Genentech, Inc. (Industry); OSI Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAO-OSI-3601S; Genentech, Inc.
Record Dates: First submitted 2006-03-16; First posted 2006-03-17 (Estimated); Results first posted 2017-07-27 (Actual); Last update posted 2017-07-27 (Actual); Status verified 2017-06

CONDITIONS: Head and Neck Cancer
Keywords: Head and Neck Cancer; Erlotinib; RADPLAT
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Erlotinib Hydrochloride; Cisplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RADPLAT and Tarceva (Experimental): All patients will receive RADPLAT and Tarceva:
  Drug: Erlotinib (Tarceva)
  150 mg daily X 7 weeks
  Other Names:
  Tarceva
  Drug: Intra-arterial Cisplatin (PLAT)
  1 dose (150 mg/sq) per week X 4 weeks
  Other Names:
  Cisplatin
  Radiation: Radiation Therapy (RAD)
  5 days per week X 7 weeks
  Interventions: Drug: Erlotinib (Tarceva); Drug: Intra-arterial Cisplatin (PLAT); Radiation: Radiation Therapy (RAD)

INTERVENTIONS:
Drug: Erlotinib (Tarceva) — 150 mg daily X 7 weeks
  Other Names: Tarceva
Drug: Intra-arterial Cisplatin (PLAT) — 1 dose (150 mg/sq) per week X 4 weeks
  Other Names: Cisplatin
Radiation: Radiation Therapy (RAD) — 5 days per week X 7 weeks

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of treatment with Tarceva (Erlotinib) and RADPLAT (RADiation and intraarterial cisPLATin) for patients with Head and Neck cancer

DETAILED DESCRIPTION:
Head and neck malignancies represent a group of epidermoid tumors that arise from the epithelial lining of the mouth, pharynx, and larynx. Three modalities of therapy have established roles in the treatment of carcinoma of the head and neck: chemotherapy, radiation therapy (XRT), and surgery. The choice of modality depends upon many factors such as the site and extent of the primary lesion, the likelihood of complete surgical resection, the presence of lymph node metastases, etc. Traditionally, smaller lesions (stage T1-T2) are effectively treated either, by surgical excision or irradiation whereas more advanced disease (stage III-IV) is treated with combined surgery and XRT. The subsequent morbidity related to extensive surgery is a major problem among survivors. Clearly, there is a need to develop therapeutic strategies for patients with advanced head and neck cancer with more effective approaches employing non-surgical modalities.

Our hypothesis is that head and neck cancers are resistant to apoptosis from DNA damage induced by radiation and chemotherapy. This resistance is mediated by EGFR overexpression which results in downstream activation of cell survival signals, such as AKT, and may be overcome when Erlotinib (Tarceva) is co-administered with RADiation and cisPLATin (intraarterial chemotherapy).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed Stage III-IV disease comprised of T3 or T4 N0-2 lesions of the oral cavity, oropharynx, hypopharynx, and larynx.
* No previous radiation therapy or chemotherapy.
* No evidence of distant metastatic disease.
* Age > 18.
* Karnofsky performance status of > 60 (ECOG 2).
* ANC > 1000, platelets > 100,000, calculated or 24-hour creatinine clearance > 60.
* Study-specific informed consent form.
* Protocol treatment must begin < 8 weeks of diagnostic biopsy.
* Ability to understand and the willingness to sign a written informed consent document.
* Patients with surgically cured secondary malignancy who have been disease free > 5 years are eligible.

Exclusion Criteria:

* Radiologic evidence of bone destruction.
* Previous or concurrent head and neck primaries.
* Prior surgery to study site other than biopsy.
* Patients receiving any other investigational agents.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to agents used in the study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because treatments and agents have the potential for teratogenic or abortifacient effects. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* History of a prior or concomitant malignancy (other than carcinoma in situ of the cervix, basal cell or squamous cell carcinoma of the skin).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2006-03; Primary Completion 2015-05 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Krishna Rao, MD, PhD, Principal Investigator — SIU School of Medicine; Thomas Robbins, MD, Principal Investigator — Simmons Cancer Institute at SIU
Locations (1):
- Simmons Cooper Cancer Institute/SIU School of Medicine, Springfield, Illinois, United States

REFERENCES:
- See also: official website of the SimmonsCooper Cancer Institute at SIU — http://www.siumed.edu/cancer/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment open between May 2006 and October 2009 at a small academic center outpatient otolaryngology/ oncology clinic.
Groups:
- RADPLAT and Tarceva: All patients will receive RADPLAT and Tarceva:
  Drug: Erlotinib (Tarceva)
  150 mg daily X 7 weeks
  Other Names:
  Tarceva
  Drug: Intra-arterial Cisplatin (PLAT)
  1 dose (150 mg/sq) per week X 4 weeks
  Other Names:
  Cisplatin
  Radiation: Radiation Therapy (RAD)
  5 days per week X 7 weeks
  Erlotinib (Tarceva): 150 mg daily X 7 weeks
  Intra-arterial Cisplatin (PLAT): 1 dose (150 mg/sq) per week X 4 weeks
  Radiation Therapy (RAD): 5 days per week X 7 weeks
Period: Overall Study
Arm/Group | RADPLAT and Tarceva
Started | 21
Completed | 19
Not Completed | 2
Not completed — lack of insurance coverage for chemoRT | 1
Not completed — PT had medical condition preventing TX | 1

BASELINE CHARACTERISTICS:
Arm/Group | RADPLAT and Tarceva
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 21
T stage of Tumor at diagnosis [Count of Participants; unit: Participants]
  T4 stage of tumor | 13
  T3 stage of tumor | 8
N stage of Tumor at diagnosis [Count of Participants; unit: Participants] — T3 Tumor > 4cm in greatest dimension
  T4a - Moderately advanced local disease
  T4b - Very Advanced local disease
  N0-no regional lymph node metastasis
  N1-metastasis in a single ipsilateral lymph node 3cm or less in greatest dimension
  N2-metastasis in a single ipsilateral lymph node > 3cm but not more than 6cm in greatest dimension; or in multiple ipsilateral lymph nodes, none > 6 cm in greatest dimension; or in bilateral or contralateral lymph nodes, none> 6 cm in greatest dimension
  N3 Metastasis in a lymph node > 6cm greatest dimension
  Participants
    N0 stage of tumor | 4
    N1 stage of tumor | 4
    N2 Stage of tumor | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete and Partial Response Using RECIST Criteria
Description: Complete and Partial Response as defined by RECIST 1.0. Complete Response (CR): Disappearance of all target lesions Partial Response (PR): At least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD
Time Frame: 17 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | RADPLAT and Tarceva
Number analyzed (Participants) | 19
Participants
  Complete Response | 17
  Partial Response | 2

2. Secondary Outcome: Survival Post Treatment
Description: Overall Survival with a minimum follow up of 1year. Relapse/Persistent Disease Rates
Time Frame: 22 months
Measure: Number; unit: participants
Arm/Group | RADPLAT and Tarceva
Number analyzed (Participants) | 19
participants | 12

ADVERSE EVENTS:
Arm/Group | RADPLAT and Tarceva
Serious Adverse Events (participants affected / at risk) | 11/19
Other Adverse Events (participants affected / at risk) | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RADPLAT and Tarceva (N=19)
Nausea (Gastrointestinal disorders) | 5
Diarrhea (Gastrointestinal disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 3
Weight loss (Investigations) | 2
vomiting (Gastrointestinal disorders) | 2
Fever (General disorders) | 2
Anemia (Blood and lymphatic system disorders) | 1
thrombocytopenia (Blood and lymphatic system disorders) | 1
Hypothermia (General disorders) | 1
Arterial Bleeding (Vascular disorders) | 1
Pain (General disorders) | 1
stridor (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RADPLAT and Tarceva (N=19)
Depression (Psychiatric disorders) | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Headache (Nervous system disorders) | 6
Mucositis (Respiratory, thoracic and mediastinal disorders) | 13
Neutropenia (Blood and lymphatic system disorders) | 8
Hearing loss (Ear and labyrinth disorders) | 6
Rash (Immune system disorders) | 12
Diarrhea (Gastrointestinal disorders) | 10
Nausea (Gastrointestinal disorders) | 7
Dehydration (Metabolism and nutrition disorders) | 8
Anemia (Blood and lymphatic system disorders) | 9
thrombocytopenia (Blood and lymphatic system disorders) | 9
weight loss (Investigations) | 8
hypoglycemia (Metabolism and nutrition disorders) | 3
pain (General disorders) | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes